CLINICAL TRIAL: NCT01334346
Title: An Investigation on Footwear Minimalism and Injury Risk in Runners
Brief Title: Footwear Minimalism Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Nike (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H11-00931
Record Dates: First submitted 2011-04-11; First posted 2011-04-13 (Estimated); Last update posted 2013-03-29 (Estimated); Status verified 2013-03

CONDITIONS: Healthy Runners
Keywords: Running; Footwear; Injury incidence; injury risk; pain
MeSH Terms: conditions — Pain

ARMS (3):
- Neutral Shoe (Active Comparator): Conventional, non-minimalist, footwear.
  Interventions: Other: Nike Pegasus
- Partial minimalist shoe (Experimental)
  Interventions: Other: Nike Free 3.0
- Full minimalist (Experimental)
  Interventions: Other: Vibram Five Fingers Shoe

INTERVENTIONS:
Other: Nike Pegasus — Conventional neutral supportive running footwear. Non minimalist.
  Arms: Neutral Shoe
Other: Nike Free 3.0 — Partial minimalist shoe with partially elevated heel, but with increased mid-sole flexibility.
  Arms: Partial minimalist shoe
Other: Vibram Five Fingers Shoe — Full minimalist shoe. Virtually no mid-sole, therefore no heel elevation or forefoot rockering. A proxy for a barefoot running condition.
  Arms: Full minimalist

SUMMARY:
The following study proposes to investigate the injury risk associated with the use of a new category of running footwear: the minimalist shoe. A group of experienced adult male and female runners with neutral foot types will take part in this study. All participants will be randomized to receive one of three different shoes: a full minimalist shoe (Vibram 5-Fingers), a partial minimalist shoe (Nike Free 3.0) and a conventional neutral supportive running shoe (Nike Pegasus), while training for a 10k event over a 14-week period. Outcomes to be investigated are pain, footwear perception, and number of injury events.

The hypothesizes is that participants using the minimalist footwear during their running program will experience a reduction in running related pain. A greater degree of footwear minimalism will result in a greater reduction in pain (compared to the partial minimalist shoe, Nike Free).

ELIGIBILITY:
Inclusion Criteria:

* Minimum of 5 years experience running
* Have been running on a regular basis (minimum once per week) over the past 6 months
* Able to run for 60 minutes continuously
* Can tolerate 20-40km per week in training
* Neutral foot posture according to the Foot Posture Index.

Exclusion Criteria:

* Have not experienced a running related injury requiring a stoppage of 2-weeks or more in the past 6 months
* History of surgery to their plantar fascia or Achilles tendon
* Have already been running in a minimalist shoe
* Have a diagnosis of osteoarthritis - or other degenerative musculoskeletal disorder - affecting the lower extremity
* Are currently taking analgesic medication.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 91 (Actual)
Dates: Start 2011-08; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Number of Injury Events | 12 weeks
  Number of run injury events (defined as unable to complete 3 consecutive running workouts due to running related pain). A calculation of injury incidence will be based on this number after dividing by the number of athletic exposures.

SECONDARY OUTCOMES:
Foot and Ankle Disability Index (FADI) | Week 12
Numerical Pain Scale (NPS) for Overall Running Related Pain | Week 12
Regional Specific NPS: Shin and Calf Pain | Week 12
Regional Specific NPS: Foot and Ankle Pain | 12 Week
Regional Specific NPS: Knee Pain | 12 Weeks
Regional Specific NPS: Pelvis and Groin Pain | 12 Week
Regional Specific NPS: Lower Back Pain | 12 Week

CONTACTS AND LOCATIONS:
Overall Officials: Jack Taunton, MD, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia, Vancouver, British Columbia, Canada